CLINICAL TRIAL: NCT01789060
Title: The Impact of Activated p-AKT Expression on Clinical Outcomes in Malignant Lymphoma : A Clinicopathological Study
Brief Title: p-AKT Expression on Clinical Outcomes in Malignant Lymphoma
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Other Study IDs: 2013-01-047
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Malignant Lymphoma; P13K-AKT Pathway Deregulation
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — paraffin-embedded biopsy specimen or unstained slides for immunostaining of p-AKT
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- p-AKT: p-AKT immunohistochemical staining,high p-AKT expression (upper quartile), low p-AKT expression (lower 3 quartiles)
  Interventions: Other: p-AKT immunohistochemical staining

INTERVENTIONS:
Other: p-AKT immunohistochemical staining — p-AKT staining on the adequate paraffin-embedded biopsy specimen or unstained slides

SUMMARY:
PI3K(phosphatidylinositol 3-kinase)/AKT pathway is an important oncogenic signaling pathway. However, clinical information about the significance of p-AKT expression in malignant lymphoma is not fully understood yet. In this study, we investigated the overexpression of p-AKT and its prognostic implication in malignant lymphoma.

DETAILED DESCRIPTION:
Recently, among diverse oncogenic signaling pathways, a number of studies have focused on the significance of oncogenic PI3K/AKT (phophatidylinositol 3-kinase/serine-threonine kinase, also known as protein kinase B [PKB]) pathway. PI3K(phosphatidylinositol 3-kinase)/AKT pathway phosphorylates and activates AKT as phosphorylated AKT (p-AKT) and plays a critical role promoting malignant phenotype and has prognostic significance in various solid cancers.

However, a systematic approach on the impact of p-AKT overexpression on clinical outcomes has not been performed in malignant lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. the patients were pathologically confirmed of malignant lymphoma, according to the World Health Organization classification;
2. the patients had adequate paraffin-embedded biopsy specimen or unstained slides for immunostaining of p-AKT.

Exclusion Criteria:

1. Primary central nervous system lymphoma was excluded in this study

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with malignant lymphoma who are treated in a tertiary hospital in Korea (Samsung Medical Center)
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Difference of overall survival according to p-AKT status in malignant lymphoma | study entry

SECONDARY OUTCOMES:
Subgroup analysis of overall survival according to histologic subtypes (GCB vs non GCB) | study entry

OTHER OUTCOMES:
Subgroup analysis of overall survival according to International Prognostic Index risk groups | study entry

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hong JY, Hong ME, Choi MK, Kim YS, Chang W, Maeng CH, Park S, Lee SJ, Do IG, Jo JS, Jung SH, Kim SJ, Ko YH, Kim WS. The impact of activated p-AKT expression on clinical outcomes in diffuse large B-cell lymphoma: a clinicopathological study of 262 cases. Ann Oncol. 2014 Jan;25(1):182-8. doi: 10.1093/annonc/mdt530. PMID 24356628